CLINICAL TRIAL: NCT00320177
Title: Eating Behavior in Children
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040050; 04-CH-0050
Record Dates: First submitted 2006-04-29; First posted 2006-05-03 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-10-28

CONDITIONS: Eating Behaviors
Keywords: Binge Eating; Food Intake; Obesity; Melanocortin-4 Receptor Gene; Child; Macronutrient Composition
MeSH Terms: conditions — Feeding Behavior; Bulimia; Obesity

SUMMARY:
This study will explore the eating habits of children and determine if eating behavior is linked to genetics.

Children between 8 and 17 years of age may be eligible for this study. It will include children who have experienced loss of control over eating, children who report overeating without loss of control, and children who report experiencing neither of the above. Candidates will be screened with the following:

* Medical history and brief physical examination, including height, weight, and body fat measurements. Body fat is measured using a device called a Bod Pod. The child sits inside the device for about 5 minutes and the machine determines body fat by measuring air movement. The child must wear a tight-fitting swimsuit for this test.
* Urine test to look for sugar or protein in the urine and to test for pregnancy in females.
* Blood tests for routine chemistries and for gene studies related to eating behaviors.
* Questionnaires and interviews about the child's general health and eating habits.
* Acclimatization to test meal conditions for the study. The child is given a yogurt shake to drink and fills out rating scales before and after the drink.

Participants will come to the Clinical Center two times at 8:30 a.m. for laboratory meal testing. At each visit, the child will do the following:

* In the morning, eat a breakfast of apple juice and a buttered English muffin.
* Between 10 a.m. and 2 p.m., pursue activities at the Clinical Center recreation facility or the NIH classroom, but may not eat or drink anything that contains calories.
* At 2 p.m., fill out rating scales about his or her hunger level.
* At 2:30 p.m., eat from a food buffet that will be made available.
* After eating, repeat rating scales about hunger level.

The procedure for both visits will be the same, except at one visit the child will be instructed to eat as much as you would eat at a normal meal, and at the other visit, the instruction will be to let yourself go and eat as much as you want.

DETAILED DESCRIPTION:
Little is known about the eating habits of children under laboratory conditions. In this exploratory study, we aim to examine the relationships between measured food intake during meals, binge eating behaviors as assessed by interview, and polymorphisms in genes believed to be involved in the regulation of energy intake. We will study children who report they have experienced loss of control over eating, children who report overeating without loss of control, and children who report neither of these episodes, and assess the impact of two different meal instructions on their eating behavior. We will ask children to eat a meal in the laboratory setting on two occasions. The only difference between the two meals will be a pre-meal instruction: Participants will be asked either to eat 'normally' (the 'normal meal' instruction) or to 'let yourself go' (the 'binge meal' instruction). Participants will be assessed for affective state; degree of hunger, fullness, and desire to binge; presence of overeating or loss of control; eating attitudes and dieting; and general school and social adjustment. Participants' DNA will be sequenced to seek polymorphisms in genes relevant for appetite, such as the leptin and melanocortin 4 receptor genes, to examine whether genetic variation in the leptin signaling pathway can account for variation in reported or actual eating behaviors. Samples will also be obtained for hormones believed to be relevant for food intake. By accurately describing eating behavior in children in relation to their age, weight, history of dieting and/or overeating behavior, and genetic variation, we can refine current theoretical models of disordered eating.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Good general health.
* Age greater than 7 and less than 18 years.
* Participants must have negative urine glucose and normal electrolytes, hepatic, and thyroid function or they will be referred for treatment.

EXCLUSION CRITERIA:

* Any major medical problem likely to affect caloric intake (e.g., significant cardiac or pulmonary disease likely to result in hypoxia or decreased perfusion).
* History of an eating disorder, other than binge eating disorder, or a current psychiatric disorder. Identification of any such illness will lead to immediate referral to a mental health professional.
* Recent weight change of greater than 5 lbs. within the previous three (3) months.
* Pregnancy. If a potential participant is found to be pregnant, we will inform the child, as an 'emancipated minor,' and let her inform her parent(s).
* Individuals who have, or whose parent or guardians have, current substance abuse or a diagnosed psychiatric disorder or other condition that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study.
* Participants currently prescribed SSRI's neuroleptics, tricyclics, stimulants, or any medication likely to affect caloric intake. Recent use (with six months) of weight loss medications.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 263 (Actual)
Dates: Start 2003-11-26; Study Completion 2014-10-28

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Spitzer RL, Yanovski S, Wadden T, Wing R, Marcus MD, Stunkard A, Devlin M, Mitchell J, Hasin D, Horne RL. Binge eating disorder: its further validation in a multisite study. Int J Eat Disord. 1993 Mar;13(2):137-53. PMID 8477283
- [Background] Smith DE, Marcus MD, Lewis CE, Fitzgibbon M, Schreiner P. Prevalence of binge eating disorder, obesity, and depression in a biracial cohort of young adults. Ann Behav Med. 1998 Summer;20(3):227-32. doi: 10.1007/BF02884965. PMID 9989331
- [Background] Striegel-Moore RH, Wilfley DE, Pike KM, Dohm FA, Fairburn CG. Recurrent binge eating in black American women. Arch Fam Med. 2000 Jan;9(1):83-7. doi: 10.1001/archfami.9.1.83. PMID 10664648
- [Derived] Manoli I, Sysol JR, Head PE, Epping MW, Gavrilova O, Crocker MK, Sloan JL, Koutsoukos SA, Wang C, Ktena YP, Mendelson S, Pass AR, Zerfas PM, Hoffmann V, Vernon HJ, Fletcher LA, Reynolds JC, Tsokos MG, Stratakis CA, Voss SD, Chen KY, Brown RJ, Hamosh A, Berry GT, Chen XS, Yanovski JA, Venditti CP. Lipodystrophy in methylmalonic acidemia associated with elevated FGF21 and abnormal methylmalonylation. JCI Insight. 2024 Feb 22;9(4):e174097. doi: 10.1172/jci.insight.174097. PMID 38271099
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281
- [Derived] Vannucci A, Tanofsky-Kraff M, Ranzenhofer LM, Kelly NR, Hannallah LM, Pickworth CK, Grygorenko MV, Brady SM, Condarco TA, Kozlosky M, Demidowich AP, Yanovski SZ, Shomaker LB, Yanovski JA. Puberty and the manifestations of loss of control eating in children and adolescents. Int J Eat Disord. 2014 Nov;47(7):738-47. doi: 10.1002/eat.22305. Epub 2014 May 30. PMID 24888295
- [Derived] Cassidy OL, Matheson B, Osborn R, Vannucci A, Kozlosky M, Shomaker LB, Yanovski SZ, Tanofsky-Kraff M. Loss of control eating in African-American and Caucasian youth. Eat Behav. 2012 Apr;13(2):174-8. doi: 10.1016/j.eatbeh.2012.01.003. Epub 2012 Jan 16. PMID 22365807
- [Derived] Shomaker LB, Tanofsky-Kraff M, Savastano DM, Kozlosky M, Columbo KM, Wolkoff LE, Zocca JM, Brady SM, Yanovski SZ, Crocker MK, Ali A, Yanovski JA. Puberty and observed energy intake: boy, can they eat! Am J Clin Nutr. 2010 Jul;92(1):123-9. doi: 10.3945/ajcn.2010.29383. Epub 2010 May 26. PMID 20504975
- [Derived] Tanofsky-Kraff M, McDuffie JR, Yanovski SZ, Kozlosky M, Schvey NA, Shomaker LB, Salaita C, Yanovski JA. Laboratory assessment of the food intake of children and adolescents with loss of control eating. Am J Clin Nutr. 2009 Mar;89(3):738-45. doi: 10.3945/ajcn.2008.26886. Epub 2009 Jan 14. PMID 19144730